CLINICAL TRIAL: NCT07028827
Title: A Phase III, Randomized, Double-blind, Multiple Doses, Placebo-controlled, Parallel-group Adaptive Study to Evaluate the Efficacy and Safety of Atropine for the Treatment of Myopia Progression in Children and Adolescents (MODERATO Study)
Brief Title: Atropine Eyedrops for Myopia Progression in Children and Adolescents (MODERATO STUDY)
Acronym: MODERATO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocus Innovation Ireland Limited (Industry)
Collaborators: Euromed Pharma Services SRL (Industry); Consorzio per Valutazioni Biologiche e Farmacologiche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCUS-Mode-CT-V1; 2023-510439-13-00 (Other: EU Clinical Trials Register); 1009562 (Other: Integrated Research Application System (IRAS)); U1111-1304-3811 (Other: WHO Universal Trial Reference Number (UTRN))
Record Dates: First submitted 2025-05-23; First posted 2025-06-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Myopia
Keywords: Myopia; Atropine sulfate; Eye drops; Short-sightedness; Eye Diseases; Paediatric population
MeSH Terms: conditions — Myopia; Eye Diseases

STUDY DESIGN:
Intervention Model Description: The study design includes 2 active arms (Atropine 0.025% or 0.05%) and a placebo arm.
  The study has a 2 stages seamless adaptive design (before/after interim analysis results). After the interim analysis, when half of the planned sample size is enrolled and the 1-year efficacy evaluation is available, the use of an adaptive trial design will be deemed:
  * each active arm will be stopped for futility if there are 8 patients or fewer (≤ 22.9%) with response (reduction in mean SE progression of at least 20% when compared with the placebo group;
  * the placebo arm will be stopped early for evidence of efficacy if there are 27 patients or more (≥ 77.1%) with response (reduction in mean SE progression of at least 20% when compared with the placebo group) in both active arms.
  Instead, if active arms show a favorable SE change but fewer than 27 responders in 1 or both active arms, an advantage for atropine can be hypothesized, allowing for sample size re-estimation to ensure adequate study power
Who Masked: Participant, Investigator
Masking Description: The study is designed as a double blinded clinical trial. During the trial, neither the participants nor the delegated staff will be aware of the group allocation. The 0.025% or 0.05% atropine eye drops and placebo eye drops will be prepared in a manner that will appear similar in appearance. The assignment of groups will not be disclosed to the subjects and the Investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): This group (N = 78 subjects) will be treated with 0.05% atropine eye drops
  Interventions: Drug: 0.05% atropine eye drops
- Group 2 (Experimental): This group (N = 78 subjects) will be treated with 0.025% atropine eye drops
  Interventions: Drug: 0.025% atropine eye drops
- Group 3 (Placebo Comparator): This group (N = 78 subjects) will be treated with placebo eye drops
  Interventions: Drug: placebo eye drops

INTERVENTIONS:
Drug: 0.05% atropine eye drops — One drop of 0.05% atropine in each eye once a day before bedtime
  Other Names: atropine sulfate eye drops solutions (0.05%)
  Arms: Group 1
Drug: 0.025% atropine eye drops — One drop of 0.025% atropine in each eye once a day before bedtime
  Other Names: atropine sulfate eye drops solutions (0.025%)
  Arms: Group 2
Drug: placebo eye drops — One drop of placebo in each eye once a day before bedtime
  Other Names: Control
  Arms: Group 3

SUMMARY:
Myopia, or shortsightedness, is a multifactorial disorder, governed by environmental and genetic factors.

Myopia is the most common ocular disorder worldwide with an increasing prevalence over the past few decades and affecting the quality of life and economic health of individuals worsening socio-economic problems.

Progressive myopia is nearly exclusively a condition of childhood and adolescence, as in most young adults, myopia has stabilized.

Myopia frequently appears in childhood, with a peak incidence occurring between 8 and 10 years of age.

The most used topical pharmacological intervention for managing childhood myopia progression is atropine, a non-selective muscarinic antagonist, which has been widely used in clinical trials in concentrations ranging from 0.01% to 1.0%.

Atropine is at present the agent with the highest efficacy and optimal safety profile to reduce myopia progression in children and adolescents.

MODERATO study, a phase III, prospective, multicentric, randomized, double blind, multiple doses, placebo-controlled parallel-group, adaptive study, aims to evaluate the efficacy and safety of 0.025% and 0.05% atropine eye drops in children and adolescents aged 3 to under 18 years old over a 24-month period, to understand its ability to manage and stop myopia getting worse. It will be conducted in 11 centers in Italy, Spain, Poland, the UK and Albania.

DETAILED DESCRIPTION:
The MODERATO study is a phase III, prospective, multicentric, randomized, double-blind, parallel group, adaptive, placebo-controlled trial. The study will be conducted in primary care and hospital settings in 3 European countries (Italy, Spain, Poland), in the UK and in Albania, involving a total of 11 centers.

The study hypothesis is that low dose (0.025% and 0.05%) of atropine eye drops will reduce the myopia progression in children and adolescents (3-18 years of age) compared with placebo eye drops, over 24 months.

A total of 234 participants from 5 countries will be estimated to take part in the study.

Eligible participants with myopia with a spherical equivalent refraction of both eyes at least -0.75 D at baseline will be randomized to treatment (0.025% atropine eye drops, 0.05% atropine eye drops) and placebo groups in 1:1:1 ratio. Each arm will consist of at least 78 individuals.

In this study, the primary objective is to evaluate efficacy of 0.025% and 0.05% atropine eye drops in children and adolescents over 24 months to slow the progression of myopia.

A formal interim efficacy analysis on the primary endpoint will be planned when the 50% of the total planned sample size has completed the 1-year treatment follow-up (105 evaluable patients in total: 35 in each arm).

"EARLY ESCAPE" Phase of Patients after Six Months of Atropine Eye Drops Treatment At the sixth month of treatment, if the patients who received the placebo treatment show worsening of their myopia, they will be switched to the active treatment. This approach is called "early escape", which ensures that the patients receive the best treatment as soon as possible, reducing the time during which they may receive ineffective treatment. The analysis will be conducted by a team of experts, Data Safety Monitoring Committee (DSMC). The treatment after the early escape will be carried out as open label study. Blinding will be maintained for the patients who do not early escape.

Analysis after One Year of Treatment When half of the patients in our study complete one year of treatment, a comprehensive analysis will be conducted to assess the effectiveness of the main treatment. This means that the results will be considered when data from 105 patients have been collected (35 in each group).

The Bayesian inference statistical technique will be used to combine and adapt the data collected during the treatment monitoring period.

Adaptive Approach

The study has been designed adaptively, which means that it can be adjusted based on the intermediate results emerging during the research. The central advantage of the adaptive design is the ability to include prospectively planned opportunities for modifying study design elements and hypotheses based upon interim data analyses. Bayesian statistics provide a method for updating information about the treatment effect as new data are observed and hence are well suited to interim analyses with accumulating efficacy data. Early stopping for statistical futility is useful in this trial as it can preserve resources that could instead be used on more promising active arms and prevent patients from being given an ineffective experimental treatment dosage. After one year of treatment, for half of the participants there are several scenarios that may occur:

1. If there are 8 or fewer people who respond positively in each group of patients who have received the active treatment (the treatment with medication), there should be the discontinuation of that treatment group as it is deemed ineffective.
2. If there are 27 or more patients who respond positively in both active treatment groups, there should be the discontinuation of the placebo treatment group, as it is confirmed that the active treatment is working well.
3. If there is a significant difference in treatment response between the active groups but the necessary number of patients to discontinue the placebo treatment arm is not reached, it could be hypothesized that the active treatment is advantageous, and the sample size of patients should be reassessed to confirm this hypothesis.

After the End of Study visit, no Follow-Up visits are foreseen. The following assessments will be performed throughout the conduction of study: Refraction test for measuring visual acuity (VA) (near and distance); Pupil diameter (PD) in photopic lighting conditions; Accommodation amplitude; Intraocular Pressure Measurement; Stereopsis; Slit lamp examination; Macular/optic disc examination by age appropriate methods (e.g. fundoscopy, or fundus photo); Ocular biometry; Instillation of cycloplegic agents, different participating site will follow their standard cycloplegic regimen (1% Tropicamide and 1% cyclopentolate eye drop); Cycloplegic autorefraction (to evaluate the refractive power of the eye); Measurement of prescription in current glasses (focimetry); Urine pregnancy test; Adverse event (AE)/Serious Adverse Event (SAE) assessments; Questionnaires (Student Refractive Error and Eyeglasses Questionnaire - Revised (SREEQ-R), Visual Light Sensitivity Questionnaire-8 (VLSQ-8), 3-items questionnaire for acceptability of the formulation) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged from 3 to less than 18 years.
* Subjects showing myopia with a spherical equivalent refraction of both eyes at least -0.75 D at baseline.
* The intraocular pressure in each eye must be equal or less than 21 mmHg.
* The parents or the legal representative must be informed about the clinical trial and must sign the informed consent form. The exception to consider is related to the individuals aged above 16 years only in the UK, who can provide their own consent according to the local regulations.
* Women with childbearing potential (WOCBP) (after menarche) who have a negative highly sensitive urine dipstick pregnancy test. Additional pregnancy testing during the study will be conducted at visits 1, 2, 3, 4, 5, 6.
* WOCBP or males who are using a highly effective birth control method to prevent pregnancies. Eligible highly effective contraceptive methods for WOCBP are combined (which contain estrogen and progestogen) hormonal contraception associated with inhibition of ovulation (oral, intravaginal (inside of the vagina), transdermal (through the skin)); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (small devices that are placed inside uterus to prevent pregnancies); intrauterine hormone-releasing system. Sexual abstinence represents a highly effective contraceptive method, if in line with the subject's normal habits.

Exclusion Criteria:

* Anisometropia, meaning a significant difference in refractive power between the two eyes exceeding |1.5| D.
* Refractive astigmatism exceeding |1.5| D.
* Presence of ocular pathologies such as pathological myopia, corneal scars, or other anterior or posterior eye pathologies.
* History of amblyopia or strabismus.
* Presence of a history of a retinal dystrophy or systemic disorder that may predispose to severe myopia (e.g., Marfan syndrome, retinitis pigmentosa, Stickler syndrome, retinopathy of prematurity)
* Abnormalities in ocular biometry, except for axial length or previous intraocular or ocular laser/non-laser surgery.
* History of glaucoma or narrow angles in the anterior chamber of the eye.
* Conditions such as Down syndrome or spastic paralysis.
* Known intolerance or allergies to atropine eye drops or hypersensitivity to any component of the atropine eye drops.
* Pregnancy or breastfeeding.
* History of alcohol or drug abuse.
* Mental or emotional instability that could interfere with study procedures.
* Lack of reliability or cooperation from the patient.
* Any treatment received for myopia within the past three months prior to inclusion in the study.
* Other reasons, at the discretion of the investigator that may deem the subject's participation in the study inappropriate.
* Patients who have consented to participate in the clinical trial, but do not meet one or more eligibility criteria required for participation in the trial during the screening procedures, and subsequently are not randomly assigned to the study treatment or entered in the study, are considered screening failures.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 234 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean annual rate of progression of myopia | 24 months
  The primary outcome measure evaluates the efficacy of atropine in slowing myopia progression in children and adolescents. The mean annual rate of progression of myopia (D/year) based on spherical equivalent (SE) measured by cycloplegic autorefraction over 24 months.

SECONDARY OUTCOMES:
Number and percentage of early escape patients. | 6 months
  To assess the early escape rate in the placebo group. Patients who show significant myopia progression at the 6-month mark will be switched to atropine eye drops at the investigator's discretion.
Mean change in axial length and glasses prescription. | 3, 6, 12, 18 and 24 months
  Assessment of the mean change in axial length (mm) and glasses prescription over a longer period of time to investigate the efficacy of the intervention.
Safety assessment of atropine. | 3, 6, 12, 18 and 24 months
  Evaluation of safety by measuring the counts and percentage of patients reporting any adverse events.
Use of photochromic and/or varifocal lenses. | 3, 6, 12, 18, and 24 months
  Number and percentage of participants requiring the use of photochromic and/or varifocal lenses.
Changes in photosensitivity index. | Baseline, 3, 6, 12, 18, and 24 months
  Evaluation of changes in photosensitivity index, used to monitor treatment-induced light sensitivity over time.
Best Corrected Visual Acuity. | 3, 6, 12, 18, and 24 months
  Assessment of best corrected distance and near visual acuity using standardised methods appropriate for participant age.
Pupil Diameter (PD) in photopic lighting condition. | 3, 6, 12, 18, and 24 months
  Measurement of PD (in mm) under photopic and average lighting using a PD ruler or autorefractor.
Accommodation amplitude. | 3, 6, 12, 18, and 24 months
  Measurement of the accommodation amplitude (diopter) performed monocularly and binocularly over distance correction.
Vision-related quality of life (SREEQ-R). | Baseline, 6, 12 and 24 months
  Patient-reported assessment of vision-related quality of life using validated questionnaire (Student Refractive Error and Eyeglasses Questionnaire - Revised - SREEQ-R) at specified time points.
Vision-related quality of life (VLSQ-8). | Baseline, 6, 12 and 24 months
  Patient-reported assessment of vision-related quality of life using validated questionnaire (Self-reported, Visual Light Sensitivity Questionnaire-8 - VLSQ-8) at specified time points.
Acceptability of atropine formulation. | 3, 6, 12, 18 and 24 months
  Assessment of acceptability of the formulation using a 3-item questionnaire, scored on a six-point scale. The questionnaire consists of a survey investigating ocular symptoms and discomforts after eye drops instillation.
Overall between-group difference from baseline in the proportion of subjects who show < -0.50 D myopia progression (Spherical Equivalent Refraction, SER). | 24 months
  Comparison of the proportion of subjects in each treatment group who show myopia progression (SER) of less than -0.50 D at 24 months. Statistical analysis will include a Chi-square test or Fisher's exact test to evaluate between-group differences.

CONTACTS AND LOCATIONS:
Overall Officials: Ian CK Wong, Professor, Principal Investigator — Ocus Innovation Ireland Limited; Annegret Dahlmann-Noor, PhD, Study Chair — NIHR Moorfields Biomedical Research Centre
Locations (11):
- University Hospital Centre Mother Teresa (UHCT), Paediatric Department, Tirana, Albania
- Italy (3):
  - Ophthalmology - AOU Consorziale Policlinico - Ospedale Pediatrico Giovanni XXIII, Bari
  - Pediatric Ophthalmology - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico Milan, Milan
  - Azienda Ospedale Università Padova, Padua
- Children's Memorial Health Institute, Department of Ophthalmology, Warsaw, Poland
- Spain (3):
  - Hospital Universitario Parc Taulí, Barcelona
  - Hospital Puerta del Mar (INIBICA), Cadiz
  - Hospital Universitario La Paz, Madrid
- United Kingdom (3):
  - Northern Ireland Clinical Research Facility. U Floor. Belfast City Hospital, Belfast
  - School of Optometry, Aston University, Birmingham
  - R&D, Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No